CLINICAL TRIAL: NCT00567996
Title: A 26-week Treatment, Multi-center, Randomized, Double-blind, Double- Dummy, Placebo-controlled, Parallel-group Study to Assess the Efficacy, and Safety of Indacaterol (150 µg o.d.) in Patients With Chronic Obstructive Pulmonary Disease, Using Salmeterol (50 µg b.i.d.) as an Active Control
Brief Title: Efficacy and Safety of Indacaterol in Patients With Chronic Obstructive Pulmonary Disease (COPD) Using Salmeterol as Active Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External affairs, novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAB149B2336
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease, indacaterol, salmeterol, placebo controlled
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Indacaterol 150 μg (Experimental): Indacaterol 150 μg once daily in the morning, inhaled via a single dose dry powder inhaler (SDDPI). Placebo to Salmeterol delivered twice daily via a proprietary dry powder inhaler in the morning and in the evening.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Placebo to Salmeterol
- Placebo (Placebo Comparator): Placebo to Indacaterol once daily in the morning, inhaled via a single dose dry powder inhaler (SDDPI). Placebo to Salmeterol delivered twice daily via a proprietary dry powder inhaler in the morning and in the evening.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Salmeterol 50 μg (Active Comparator): Salmeterol 50 μg twice daily delivered via a proprietary dry powder inhaler in the morning and in the evening. Placebo to Indacaterol daily in the morning, inhaled via a single dose dry powder inhaler (SDDPI).
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Salmeterol 50 μg; Drug: Placebo to Indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol 150 μg once daily (o.d) inhaled
  Arms: Indacaterol 150 μg
Drug: Salmeterol 50 μg — Salmeterol 50 μg twice daily (b.i.d) delivered via a proprietary dry powder inhaler
  Arms: Salmeterol 50 μg
Drug: Placebo to Indacaterol — Placebo to Indacaterol inhaled via SDDPI.
  Arms: Placebo; Salmeterol 50 μg
Drug: Placebo to Salmeterol — Placebo to salmeterol delivered via a proprietary dry powder inhaler
  Arms: Indacaterol 150 μg; Placebo

SUMMARY:
This study evaluated the safety and efficacy of 26 weeks treatment with indacaterol, placebo or salmeterol in patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of moderate to severe Chronic Obstructive Pulmonary Disease (COPD) as per the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2006 Guidelines (mandatory) and including:

* Smoking history of at least 20 pack years
* Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) < 80% predicted and >or= 30% of predicted normal value
* Post-bronchodilator FEV1/FVC < 70%

("Post" defined as within 30 minutes of inhalation of 400 µg salbutamol)

Exclusion Criteria:

* Pregnant or nursing (lactating) women and women of child-bearing potential UNLESS they meet pre-specified definitions of post-menopausal or are using pre-specified acceptable methods of contraception
* Hospitalisation for COPD exacerbation in the 6 weeks prior to Visit 1 or during run-in
* Patients requiring oxygen therapy for chronic hypoxemia (typically >15h/day)
* Respiratory tract infection within 6 weeks prior to Visit 1 and during the run-in period
* Concomitant pulmonary disease
* Asthma history (eosinophils > 400/mm3; symptoms prior to age 40). Includes history of childhood asthma
* History of long QTc syndrome or QTc interval > 450 ms for males and >470 ms for females
* Patients who have a clinically significant condition or a clinically relevant laboratory abnormality
* History of reactions to sympathomimetic amines or inhaled medication
* Inability to use the dry powder devices or perform spirometry
* Irregular day/night, wake/sleep cycles, e.g. shift workers
* Certain medications for COPD and allied conditions such as long acting bronchodilators must not be used prior to Visit 1 and for a pre-specified minimum washout period
* Patients unable or unwilling to complete a patient diary

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (127):
- Canada (6):
  - Novartis Investigative Site, Edmonton
  - Novartis Investigator Site, Edmonton
  - Novartis Investigator Site, London
  - Novartis Investigator Site, Mirabel
  - Novartis Investigator Site, Montreal
  - Novartis Investigator Site, Toronto
- Colombia (3):
  - Novartis Investigator site, Barranquilla
  - Novartis Investigator Site, Bogota D.C.
  - Novartis Investigator Site, Medellín
- Czechia (6):
  - Novartis Investigator Site, Cvikov
  - Novartis Investigator Site, Lovosice
  - novartis Investigator site, Novy Jocin
  - Novartis Investigator Site, Pardubice
  - Novartis Investigator Site, Prague
  - Novartis Investigative Site, Žatec
- Denmark (12):
  - Novartis Investigator Site, Aalborg
  - Novartis Investigator Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigator Site, Copenhagen
  - Novartis Investigator Site, Frederikssund
  - Novartis investigator site, Hellerup
  - Novartis Investigator site, Hvidovre
  - Novartis investigator site, Odense
  - Novartis Investigator Site, Roslev
  - Novartis Investigative Site, Silkeborg
  - Novartis Investgative Site, Søborg
  - Novartis Investigator Site, Vaerloese
- Finland (6):
  - Novartis Investigator Site, Hus
  - Novartis Investigator Site, Jyväskylä
  - Novartis Investigator Site, Lahti
  - Novartis Investigator Site, Oulu
  - Novartis Investigator Site, Tampere
  - Novartis Investigator Site, Turku
- France (4):
  - Novartis Investigative Site, Ambroise
  - Novartis Investigative Site, Beuvry
  - Novartis Investgative Site, Férolles-Attilly
  - Novartis Investigator Site, Nice
- Germany (37):
  - Novartis Investigator Site, Bad Segeberg
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bielefeld
  - Novartis Investigator Site, Bochum
  - Novartis Investigator Site, Bonn
  - Novartis Investigator Site, Brühl
  - Novartis Investigator Site, Cologne
  - Novartis Investigator Site, Cottbus
  - Novartis Investigator Site, Dortmund
  - Novartis Investigator Site, Düren
  - Novartis Investigator Site, Eggenfelden
  - Novartis investigator site, Eschwege
  - Novartis Investigator Site, Forchheim
  - Novartis Investigator Site, Freudenberg
  - Novartis Investigator Site, Fürth
  - Novartis Investigator Site, Gelsenkirchen
  - Novartis Investigator Site, Gummersbach
  - Novartis Investigator Site, Hagen
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Kassel
  - Novartis Investigator Site, Kempten
  - Novartis Investigator Site, Landsberg am Lech
  - Novartis Investigator Site, Langenfeld
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Munich
  - Novartis Investigator Site, München
  - Novartis Investigator Site, Neuss
  - Novartis Investigator Site, Nuremberg
  - Novartis Investigator Site, Oschersleben
  - Novartis Investigator Site, Ruhmannsfelden
  - Novartis Investigator site, Sinsheim
  - Novartis Investigator Site, Solingen
  - Novartis Investigator Site, Steinfort-borghorst
  - Novartis Investigator Site, Vilshofen
  - Novartis Investigator Site, Wallerfing
  - Novartis Investigator Site, Witten
- Hungary (5):
  - Novartis Investigator Site, Budapest
  - Novartis investigator site, Debrechen
  - Novartis Investigator Site, Deszk
  - Novartis Investigator Site, Mosonmagyaróvár
  - Novartis Investigator Site, Székesfehérvár
- Novartis investigator site, Reykhavik, Iceland
- India (9):
  - Novartis Investigator Site, Chennai
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigator Site, Goa
  - Novartis Investigator Site, Hyderabad
  - Novartis Investigator Site, Jaipur
  - Novartis Investigator Site, Kerala
  - Novartis Investigator Site, Mangalore
  - Novartis Investigator Site, Mumbai
  - Novartis Investigator Site, Vellore
- Italy (15):
  - Novartis Investigator Site, Ancona
  - Novartis Investigator Site, Arenzano
  - Novartis Investigative Site, Ascoli Piceno
  - Novartis Investigator Site, Brescia
  - Novartis Investigator Site, Cagliari
  - Novartis investigator site, Chieti
  - Novartis Investigator Site, Ferrara
  - Novartis Investigator Site, Milan
  - Novartis Investigator Site, Orbassano
  - Novartis Investigator Site, Palermo
  - Novartis Investigator Site, Reggio Emilia
  - Novartis Investigator Site, Rome
  - Novartis Investigator Site, Sexten
  - Novartis Investigator Site, Siena
  - Novartis Investigator Site, Terni
- Peru (6):
  - Novartis Investigator Site, Callao
  - Novartis Investigator Site, Miraflores
  - Novartis Investigator Site, San Borja
  - Novartis Investigator Site, San Isidro
  - Novartis Investigator Site, San Martín de Porres
  - Novartis Investigator Site, Surco
- Russia (6):
  - Novartis Investigator Site, Kazan'
  - Novartis Investigator Site, Moscow
  - Novartis Investigator Site, Saint Petersburg
  - Novartis Investigator Site, Samara
  - Novartis Investigator Site, Yaroslavl
  - Novartis Investigator Site, Yekaterinburg
- Slovakia (5):
  - Novartis Investigator Site, Bardejov
  - Novartis Investigator Site, Bratislava
  - Novartis Investigator Site, Košice
  - Novartis Investigator Site, Kovice
  - Novartis Investigator Site, Spišská Nová Ves
- Taiwan (6):
  - Novartis Investigator Site, Changhua
  - Novartis Investigator Site, Kaohsiung City
  - Novartis Investigator Site, Kaohusing
  - Novartis Investigator Site, Lin-ko
  - Novartis Investigator Site, Taichung
  - Novartis Investigator Site, Taipei

REFERENCES:
- [Derived] Yelensky R, Li Y, Lewitzky S, Leroy E, Hurwitz C, Rodman D, Trifilieff A, Paulding CA. A pharmacogenetic study of ADRB2 polymorphisms and indacaterol response in COPD patients. Pharmacogenomics J. 2012 Dec;12(6):484-8. doi: 10.1038/tpj.2011.54. Epub 2011 Dec 13. PMID 22158330
- [Derived] Jones PW, Mahler DA, Gale R, Owen R, Kramer B. Profiling the effects of indacaterol on dyspnoea and health status in patients with COPD. Respir Med. 2011 Jun;105(6):892-9. doi: 10.1016/j.rmed.2011.02.013. Epub 2011 Mar 11. PMID 21397482
- [Derived] Worth H, Chung KF, Felser JM, Hu H, Rueegg P. Cardio- and cerebrovascular safety of indacaterol vs formoterol, salmeterol, tiotropium and placebo in COPD. Respir Med. 2011 Apr;105(4):571-9. doi: 10.1016/j.rmed.2010.11.027. Epub 2011 Jan 11. PMID 21227674

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1002 participants were randomized. 3 randomized participants in the Indacaterol group and 1 randomized participant in the Salmeterol group did not receive study medication and were not included in the intent-to-treat milestone.
Groups:
- Placebo: Placebo to indacaterol inhaled via SDDPI. Placebo to salmeterol delivered twice daily via a proprietary dry powder inhaler in the morning and in the evening. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
Period: Overall Study
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Started | 333 (Randomized participants) | 334 | 335
Intent-to-treat: Received Study Drug | 330 | 333 | 335
Completed | 289 | 284 | 265
Not Completed | 44 | 50 | 70
Not completed — Adverse Event | 18 | 16 | 13
Not completed — Protocol Deviation | 9 | 11 | 13
Not completed — Withdrawal by Subject | 8 | 12 | 22
Not completed — Abnormal Lab value(s) | 2 | 1 | 2
Not completed — Abnormal test procedure result(s) | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 5 | 2
Not completed — Unsatisfactory therapeutic effect | 1 | 2 | 15
Not completed — Administrative problems | 1 | 1 | 0
Not completed — Death | 1 | 0 | 2
Not completed — Patient's inability to use the device | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Placebo | Total
Number analyzed (Participants) | 330 | 333 | 335 | 998
Age Continuous [Mean (Standard Deviation); unit: years] — All baseline measures are based on the intent-to-treat population that included all randomized participants who received at least one dose of study medication.
  years | 63.2 (8.67) | 63.4 (9.19) | 63.9 (8.56) | 63.5 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 84 | 77 | 253
  Male | 238 | 249 | 258 | 745

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 12 Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 hour 10 minute and 23 hour 45 minute post-dose FEV1 readings. Mixed model used baseline FEV1, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, and FEV1 prior to and 1 hour post inhalation of ipratropium as covariates.
Time Frame: Week 12
Population: Intent-to-treat population included all randomized participants who received at least one dose of study medication. The end point was analyzed only for those participants who had Trough FEV1 data at week 12. Missing data were imputed using Last Observation carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Number analyzed (Participants) | 320 | 317 | 316
Liters | 1.45 (0.018) | 1.39 (0.018) | 1.28 (0.019)

2. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score After 12 Weeks of Treatment
Description: SGRQ is a health related quality of life questionnaire consisting of 76 items in three sections: symptoms, activity and impacts. The total score is 0 to 100 with a higher score indicating poorer health status. The mixed model used baseline SGRQ total score, FEV1 prior to and 30 minutes post inhalation of salbutamol/albuterol, and FEV1 prior to and one hour post inhalation of ipratropium as covariates.
Time Frame: Week 12
Population: Intent-to-treat population included all randomized participants who received at least one dose of study medication. The endpoint was analyzed only for those participants who had SGRQ data at week 12. Missing data were imputed using Last Observation carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Number analyzed (Participants) | 309 | 301 | 294
Score on a scale | 36.4 (1.04) | 38.5 (1.04) | 42.6 (1.05)

3. Secondary Outcome: Percentage of COPD "Days of Poor Control" During 26 Weeks of Treatment
Description: Participants rated their symptoms on a scale of 0=none to 3=severe. A Chronic Obstructive Pulmonary Disease (COPD) "day of poor control" was defined as any day in the participants diary with a score >=2 (moderate or severe) for at least 2 of 5 symptoms (cough, wheeze, production of sputum, color of sputum, breathlessness). The mixed model used baseline percentage of "days of poor control", FEV1 prior to and 30 minutes post inhalation of salbutamol/albuterol, and FEV1 prior to and one hour post inhalation of ipratropium as covariates.
Time Frame: Up to 26 weeks
Population: Intent-to-treat population included all randomized participants who received at least one dose of study medication. The endpoint was analyzed only for those participants who had data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Number analyzed (Participants) | 310 | 310 | 304
Percentage of days | 34.1 (1.82) | 34.1 (1.82) | 38.1 (1.85)

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Safety population consisting of all participants who received at least one dose of study medication.
Arm/Group | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 29/330 | 19/333 | 26/335
Other Adverse Events (participants affected / at risk) | 69/330 | 68/333 | 71/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=330) | Salmeterol 50 μg (N=333) | Placebo (N=335)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cor pulmonale acute (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 3 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 2 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=330) | Salmeterol 50 μg (N=333) | Placebo (N=335)
Nasopharyngitis (Infections and infestations) | 24 | 29 | 21
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 52 | 48 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. any publications from a single-site are postponed until the publication of the pooled date (i.e., data from all sites) in the clinical trial.